CLINICAL TRIAL: NCT03396289
Title: The Effects of Balance and Respiratory Muscle Training on Functional Capacity, Balance, Respiratory Function and Respiratory Muscle Strength in Children With Cerebral Palsy
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: Bezmialem Vakif University (Other)
Responsible Party: Principal Investigator, Büşra Kepenek Varol, Lecturer, PT, MSc, Bezmialem Vakif University
Allocation: Randomized | Model: Parallel | Masking: Double | Purpose: Treatment
Other Study IDs: bvubkvarol01
Record Dates: First submitted 2018-01-05; First posted 2018-01-10 (Actual); Last update posted 2018-06-28 (Actual); Status verified 2018-06

CONDITIONS: Cerebral Palsy, Spastic
Keywords: Cerebral Palsy; Balance; Inspiratory Muscle Training; 6-Minute Walk Test; Pulmonary Function Test; Postural Stability
MeSH Terms: conditions — Cerebral Palsy

STUDY DESIGN:
Who Masked: Participant, Outcomes Assessor
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (2):
- Control Group (Active Comparator): Patients in this group will receive conventional physiotherapy programme including balance exercises, 3 times a week for 8 weeks. One exercise session will be performed under the supervision of a physiotherapist, other 2 sessions will be performed at home.
  Interventions: Other: Conventional physiotherapy including balance exercises
- Training Group (Experimental): In addition to conventional physiotherapy programme, patients in this group will also receive inspiratory muscle training for 15 minutes, twice a day, 7 days a week for 8 weeks. One exercise session will be performed under the supervision of a physiotherapist, other sessions will be performed at home.
  Interventions: Other: Conventional physiotherapy including balance exercises; Other: Inspiratory muscle training

INTERVENTIONS:
Other: Conventional physiotherapy including balance exercises — Programme will include balance exercises with balance board and swiss ball, weight shifting exercises on board, one-legged balance, balance on unstable surface, balance on tilting surface and balance with Biodex Balance System. Biodex Balance System Biodex will only be used during sessions under physiotherapist supervision.
Other: Inspiratory muscle training — Threshold IMT device will be used for the training. Training intensity will set at 30% of the maximum inspiratory pressure.
  Arms: Training Group

SUMMARY:
Cerebral palsy (CP) is a permanent, non-progressive disorder in which the immature brain is affected by various causes in the prenatal, perinatal or postnatal period. Damage to the central nervous system in children with CP causes motor problems, balance and postural disorders. It is reported in the literature that the effects of balance and the effects of balance exercises in children with CP, similarly respiratory effects were also investigated. Balance and balance responses are especially important in children with ambulatory SP and balance problems are seen in most CP children. Insufficient control of respiratory muscles affects pulmonary ventilation negatively in children with CP. However, it seems that CP has limited articles in which respiratory muscle strength is investigated, and also limited studies involving inspiratory muscle training. Inspiratory muscle training is shown to improve pulmonary function and diaphragm (which is one of the core muscles) strength and have an effect on balance. Studies showed that respiratory muscle strength in children with CP is lower than in children with normal development. Nevertheless, there was no study showing the effects of respiratory muscle training on functional capacity and balance in children with CP. The aim of this study is to investigate the effects of balance training and inspiratory muscle training on functional capacity, balance, respiratory function and respiratory muscle strength in children with CP.

ELIGIBILITY:
Inclusion Criteria:

* Cerebral palsy diagnosis
* Children with level I or II according to Gross Motor Classification System

Exclusion Criteria:

* Orthopedic surgery and / or Botox application in the lower extremity in the last 6 months
* Severe convulsions that can not be controlled by drugs
* Congenital malformation accompanying cerebral palsy

Ages: 7 Years to 16 Years | Sex: All | Healthy Volunteers: No
Age Groups: Child
Enrollment: 30 (Actual)
Dates: Start 2018-02-23 (Actual); Primary Completion 2018-06-25 (Actual); Study Completion 2018-06-25 (Actual)

PRIMARY OUTCOMES:
Change from baseline maximum inspiratory pressure at 8 weeks | Eight weeks
Change from baseline maximum expiratory pressure at 8 weeks | Eight weeks
Change from baseline distance covered in six-minute walk test at 8 weeks | Eight weeks
Change from baseline Forced Vital Capacity (FVC) at 8 weeks | Eight weeks
Change from baseline Forced Expiratory Volume in 1 second (FEV1) at 8 weeks | Eight weeks
Change from baseline Peak Expiratory Flow (PEF) at 8 weeks | Eight weeks
Change from baseline postural stability test score in Biodex Balance System SD at 8 weeks | Eight weeks
Change from baseline limits of stability test score in Biodex Balance System SD at 8 weeks | Eight weeks
Change from baseline sensory integration and balance test score in Biodex Balance System SD at 8 weeks | Eight weeks

CONTACTS AND LOCATIONS:
Locations (1):
- Bezmialem Vakif University, Istanbul, Turkey (Türkiye)

IPD SHARING:
Plan to Share IPD: Undecided